CLINICAL TRIAL: NCT00301340
Title: An Open Trial to Evaluate the Efficacy and Safety of Summers Non-Pesticide Lice Asphyxiator (L.A.) for the Treatment of Head Lice
Brief Title: Efficacy and Safety of Summers Non-Pesticide Lice Asphyxiator (L.A.)for the Treatment of Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Summers Laboratories (Industry)
Purpose: Treatment
Other Study IDs: SU-03-2005
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Head Lice

INTERVENTIONS:
Drug: 5% Lice Asphyxiator lotion - Summers Laboratories, Inc.

SUMMARY:
Summers Laboratories has developed a non-pesticide treatment for head lice. Lice Asphyxiator (L.A.) works by mechanically blocking the respiratory spiracles of the head lice, therefore causing a quick-acting suffocation that will not result in the development of resistance.

The objectives of this open label study are to evaluate the efficacy and safety of home use of two 10-minute treatments of 5% L.A. (applied one week apart).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 6 months of age or older.
2. Have an active infestation with Pediculus capitis, the human head louse, with at least three live lice at baseline, or treatment failure with any live lice from Protocol SU-01-2005 or Protocol SU-02-2005.
3. Agree not to use any other pediculicides or medicated hair grooming products during the duration of the study.
4. Be healthy, non-febrile, and not suffering from an infection likely to require antibiotic therapy during the study period.
5. Subject or guardian is able to understand the new HIPAA regulations and sign the HIPAA form.
6. Subject or guardian has read, understood, and signed appropriate informed consent in English. If English is not the primary language, the information about the study must be explained in their language and a copy of the informed consent must be in that language.
7. Subject is willing to participate in the study, and abide by the protocol requirements.

   -

Exclusion Criteria:

1. Participation in any clinical study, excluding protocols SU-01-2005 and SU-02-2005, within the past 30 days.
2. Known hypersensitivity to any ingredient in the product formulation.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Terri Meinking, Principal Investigator — Global Health Association of Miami; Anne Lucky, Dr., Principal Investigator — Dermatology Research Associates; Jon Thomas, Dr., Principal Investigator — Alegent Health; E.A. Clark, Dr., Principal Investigator — Diagnostic Clinic of Longview, Tx; Peter E Silas, Dr., Principal Investigator — Advanced Clinical Research Institute
Locations (5):
- United States (5):
  - Global Health Associates of Miami 7800, SW 57 Avenue, Suite 219E, Miami, Florida
  - Alegent Health, Harmony Street, 2nd Floor, Council Bluffs, Iowa
  - Dermatology Research Associates 7691 Five Mile Road, Suite 312, Cincinnati, Ohio
  - Diagnostic Clinic of Longview, TX 707 Hollybrook Drive, Longview, Texas
  - Wee Care Pediatrics, 1580 West Antelope Drive, Suite 100, Layton, Utah

REFERENCES:
- [Derived] Meinking TL, Villar ME, Vicaria M, Eyerdam DH, Paquet D, Mertz-Rivera K, Rivera HF, Hiriart J, Reyna S. The clinical trials supporting benzyl alcohol lotion 5% (Ulesfia): a safe and effective topical treatment for head lice (pediculosis humanus capitis). Pediatr Dermatol. 2010 Jan-Feb;27(1):19-24. doi: 10.1111/j.1525-1470.2009.01059.x. PMID 20199404
- See also: Related Info — http://www.sumlab.com